CLINICAL TRIAL: NCT04877821
Title: An Open-label Phase II Trial Evaluating the Efficacy and Safety of Sintilimab Plus Anlotinib Combined With Chemotherapy as Neoadjuvant Therapy in Early-stage Triple-negative Breast Cancer（NeoSACT）
Brief Title: The Efficacy and Safety of Sintilimab Plus Anlotinib Combined With Chemotherapy as Neoadjuvant Therapy in TNBC
Acronym: NeoSACT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, Clinical Professor, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-19
Record Dates: First submitted 2021-04-30; First posted 2021-05-07 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Triple Negative Breast Cancer
Keywords: TNBC; neoadjuvant; immunotherapy; anti-angiogenesis
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sintilimab; anlotinib; Taxes; Carboplatin; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Patient enrollment followed a Simon two-stage design.The Simon design required 11 patients for the first stage and called for termination at stage 1 if there were less than 5 responders (Pathological complete response, pCR) among 11 patients. Otherwise, if seven or more responders were identified in up to 11 patients, additional 20 patients would be enrolled. Treatment was considered of clinical interest if, at the end of the second stage, there were more than 16 responders among 31 patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sintilimab + Anlotinib + Chemotherapy (Experimental): Experimental: Sintilimab + Anlotinib + Chemotherapy Participants receive Sintilimab every 3 weeks (Q3W) + Anlotinib d1-14 (Q3W) + (Nab paclitaxel weekly + carboplatin (Q3W) x 4 cycles followed by epirubicin + cyclophosphamide Q3W x 4 cycles) as neoadjuvant therapy prior to surgery. After surgery, the subjects will continue to receive sintilimab treatment until one year has elapsed since the start of neoadjuvant therapy (that is, they will receive sintilimab treatment at least 17 times).
  Interventions: Drug: Sintilimab; Drug: Anlotinib; Drug: Nab paclitaxel; Drug: Carboplatin; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Sintilimab — 200mg on days 1 (Q3W) of the neoadjuvant and adjuvant phase of the study; IV injection.
Drug: Anlotinib — 12mg on d1-14 of Cycles 1-8 (Q3W) of the neoadjuvant phase of the study; po. Arotinib is a small molecule multi-target TKI, which exerts its effect by inhibiting angiogenesis, a critical component of tumour growth and metastasis.
Drug: Nab paclitaxel — 100 mg/m² on day 1, 8 and 15 of Cycles 1-4 (Q3W) of the neoadjuvant phase of the study; IV injection.
Drug: Carboplatin — AUC 5 on days 1 of Cycles 1-4 (Q3W) of the neoadjuvant phase of the study; IV injection.
Drug: Epirubicin — 90 mg/m² on day of Cycles 5-8 (Q3W) of the neoadjuvant phase of the study; IV injection.
Drug: Cyclophosphamide — 600 mg/m² on day of Cycles 5-8 (Q3W) of the neoadjuvant phase of the study; IV injection.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Sintilimab plus anlotinib combined with chemotherapy as neoadjuvant therapy in participants who have triple negative breast cancer (TNBC). After a screening phase of approximately 28 days, each participant will receive neoadjuvant study treatment (Sintilimab + anlotinib + chemotherapy) based on schedule for approximately 24 weeks (8 cycles). Each participant will then undergo definitive surgery 4-6 weeks after conclusion of the last cycle of the neoadjuvant study treatment. Following adjuvant study treatment, each participant will be monitored for safety, survival and disease recurrence. The primary outcome measure is pathological complete response (pCR) rate using the definition of ypT0/Tis ypN0.

ELIGIBILITY:
Inclusion Criteria:

* Has newly diagnosed, locally advanced TNBC, as defined by the most recent American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines.
* Has previously untreated locally advanced non-metastatic (M0) TNBC defined as the following combined primary tumor (T) and regional lymph node (N) staging per current American Joint Committee of Cancer (AJCC) staging criteria for breast cancer as assessed by the investigator based on radiological and/or clinical assessment:

T1c, N1-N2 T2, N0-N2 T3, N0-N2 T4a-d, N0-N2

* Provides a core needle biopsy consisting of at least 2 separate tumor cores from the primary tumor at screening to the central laboratory.
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 performed within 10 days of treatment initiation.
* Demonstrates adequate organ function.
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 12 months after the last dose of study treatment for participants who have received cyclophosphamide, and 6 months after the last dose of study treatment for participants who did not.

Exclusion Criteria:

* Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Has received prior chemotherapy, targeted therapy, and radiation therapy within the past 12 months.
* Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed death - ligand 1 (anti-PD-L1), or antiangiogenic drug therapy.
* Is currently participating in or has participated in an interventional clinical study with an investigational compound or device within 4 weeks of the first dose of treatment in this current study.
* Has received a live vaccine within 30 days of the first dose of study treatment.
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (i.e., dosing exceeding 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B or Hepatitis C.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has significant cardiovascular disease, such as: history of myocardial infarction, acute coronary syndrome or coronary angioplasty/stenting/bypass grafting within the last 6 months OR congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV or history of CHF NYHA Class III or IV.
* Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study, starting with the screening visit through 12 months after the last dose of study treatment for participants who have received cyclophosphamide, and for 6 months after the last dose of study treatment for participants who have not.
* Has a known hypersensitivity to the components of the study treatment or its analogs.
* Has a known history of active tuberculosis (TB, Bacillus Tuberculosis).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate using the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery | Up to approximately 30-32 weeks
  pCR rate (ypT0/Tis ypN0) is defined as the percentage of participants without residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current American Joint Committee on Cancer (AJCC) staging criteria assessed by the local pathologist at the time of definitive surgery.

SECONDARY OUTCOMES:
Residual cancer burden (RCB) | Up to approximately 30-32 weeks
  Residual cancer burden (RCB)
Event-free Survival (EFS) as assessed by Investigator | Up to approximately 3 years
  EFS is defined as the time from randomization to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause.
Overall survival (OS) | Up to approximately 5 years
  OS is defined as the time from randomization to death due to any cause.
Immune response biomarkers | Up to approximately 60 weeks
  PDL1, CD8, Tils, HRD...
Percentage of participants who experience an adverse event (AE) | Up to approximately 60 weeks
  An AE is defined as any untoward medical occurrence in a participant administered study treatment which does not necessarily have to have a causal relationship with this treatment. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment or protocol-specified procedure, whether or not considered related to study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE.

OTHER OUTCOMES:
European Orgnisation for Research and Treatment of Cancer (EORTC) Quality of Life Core 30 Questionnaire (QLQ-C30) score | Up to approximately 48-52 weeks
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Individual responses are given on a 4-point scale (1=Not at All to 4=Very Much), with a lower score indicating a better outcome.
EORTC Breast Cancer-Specific QoL Questionnaire (QLQ-BR42) score | Up to approximately 48-52 weeks
  The EORTC-QLQ-BR42 is a 42-item questionnaire developed to assess the quality of life of breast cancer patients. And it is now a fully validated EORTC questionnaire and can be used in conjunction with the QLQ-C30. Individual responses are given on a 4-point scale (1=Not at All to 4=Very Much), with a lower score indicating a better outcome.
Patient Health Questionnaire-9 (PHQ-9) | Up to approximately 48-52 weeks
  PHQ-9 is a nine-item questionnaire for screening depression symptoms and measuring its severity rated on a scale of 0 (not at all), 1 (several days), 2 (more than half the days) or 3(nearly every day). The severity of depressive symptoms in this study will be classified into three subgroups according to the PHQ-9 score: no depression (0-4), mild depression (5-9) and moderate-to-severe depression (≥10). The cutoff score and its severity of PHQ-9 had been extensively applied to screen symptoms of depression in studies involving patients with cancer.
Generalized Anxiety Disorder 7-item (GAD-7) | Up to approximately 48-52 weeks
  GAD-7 is a seven-item questionnaire for screening anxiety symptoms and measuring its severity rated on a scale of 0 (not at all), 1 (several days), 2 (more than half the days) or 3 (nearly every day). The severity of anxiety symptoms in this study will be classified into three subgroups based on the GAD-7 scores: no anxiety (0-4), mild anxiety (5-9) and moderate-to-severe anxiety(≥10).GAD-7 had shown satisfactory validity and reliability for screening anxiety symptoms with cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- NeoSACT, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Yang L, Ge Y, Zhu Z, Chen B, Yang C, Gao H, Yang M, Zhu T, Wang K. Neoadjuvant anlotinib/sintilimab plus chemotherapy in triple-negative breast cancer (NeoSACT): Phase 2 trial. Cell Rep Med. 2025 Jul 15;6(7):102193. doi: 10.1016/j.xcrm.2025.102193. Epub 2025 Jun 19. PMID 40541191